CLINICAL TRIAL: NCT05553093
Title: Nanjing First Hospital, Nanjing Medical University
Brief Title: Effects of Tirzepatide and Insulin Glargine on Glucolipid Metabolism and Brain Function in Patients With Type 2 Diabetes
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20220124-02
Record Dates: First submitted 2022-04-12; First posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Tirzepatide; Insulin Glargine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tirzepatide (Experimental): Tirzepatide 5、10、15mg
  Interventions: Drug: Tirzepatide
- Insulin Glargine (Active Comparator): Insulin Glargine 6 international unit (IU)
  Interventions: Drug: Insulin Glargine

INTERVENTIONS:
Drug: Tirzepatide — Tirzepatide ih qw
  Other Names: Tirzepatide 5、10、15mg
  Arms: Tirzepatide
Drug: Insulin Glargine — 6 IU ih qd
  Other Names: Adjust insulin dose according to fasting plasma glucose (FBG)
  Arms: Insulin Glargine

SUMMARY:
The effects of Tirzepatide and Insulin Glargine on glucose and lipid metabolism and inflammation in patients with type 2 diabetes mellitus. Effects of Tirzepatide on the occurrence and development of cognitive impairment in diabetic patients and its associated pattern of changes in brain neural network characteristics.

DETAILED DESCRIPTION:
The aim of the study is to investigate the effects of Tirzepatide and Insulin Glargine on glucose and lipid metabolism and inflammation in patients with type 2 diabetes mellitus. Meanwhile, this study will evaluate the effects of Tirzepatide on the development of cognitive impairment and its associated pattern of changes in neural network characteristics in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes was diagnosed according to World Health Organization(WHO) classification or other locally applicable diagnostic criteria.
* Received stable metformin with or without sulfonylureas at least 2 months prior to visit 1 and between visits 1 and 3 (metformin ≥ 1000 mg/ day and does not exceed the maximum dose specified in the nationally approved guidelines;Sulfonylureas should be at least half of the maximum dose as stated in the national approved instructions).
* No insulin treatment (except for gestational diabetes or short-term use in acute Settings [duration ≤14 days]).
* At visit 1, HbA1c ≥ 7.5% and ≤ 11.0% was determined according to the central laboratory.
* Body mass index (BMI) ≥ 23 kg/m2.

Exclusion Criteria:

* Type 1 Diabetes Mellitus (T1DM)
* Had chronic or acute pancreatitis at any time prior to visit 1.
* A history of proliferative diabetic retinopathy or diabetic macular degeneration or non-proliferative diabetic retinopathy requiring acute treatment.
* History of severe hypoglycemia and/or insensitive hypoglycemia within 6 months prior to visit 1.
* History of ketoacidosis or hyperosmolar state/coma
* Have a known clinically significant gastric emptying disorder (e.g., severe diabetic gastroparesis or gastric outlet obstruction), have received or plan to undergo gastric bypass surgery or restrictive bariatric surgery (e.g., Lap-Band®) during the study period, or take long-term medications that directly affect gastrointestinal motility.
* Had any of the following cardiovascular diseases in the 2 months prior to the visit: acute myocardial infarction or cerebrovascular accident (stroke) or hospitalization due to congestive heart failure (CHF).
* New York Heart Association Classification of Heart Function Class III and Class IV CHF.
* Have acute or chronic hepatitis, have signs or symptoms of any liver disease other than non-alcoholic fatty liver disease (NAFLD), or have alanine aminotransferase (ALT) levels > 3.0 times the upper limit of the normal range determined by the central laboratory at visit 1;For NAFLD patients, only ALT levels ≤ 3.0 times the upper limit of the normal range (ULN) were eligible for this trial.
* The estimated glomerular filtration rate (eGFR) calculated based on the Chronic Kidney Disease Epidemiology Collaboration equation（CKD-EPI）formula was less than 45 mL/min/1.73 m2, as determined by the central laboratory at visit 1.
* The researchers suggest that there is evidence of significant, poorly controlled endocrine abnormalities, such as thyrotoxicosis or adrenal crisis.
* Family or personal history of medullary thyroid cancer (MTC) or type 2 multiple endocrine tumor syndrome.
* Serum calcitonin level ≥ 35 ng/L (pg/mL) was determined by the central laboratory at visit 1.
* There was significant evidence of active autoimmune abnormalities (e.g., lupus or rheumatoid arthritis) and the investigators suggested that systemic glucocorticoid therapy might be required in the following 12 months.
* Has received an organ transplant (corneal transplant allowed) or is waiting for an organ transplant.
* A history of active or untreated malignancy, or a remission period of less than 5 years for a clinically significant malignancy (other than basal or squamous cell skin cancer, carcinoma in situ of the cervix, or carcinoma in situ of the prostate).
* Presence of any other medical history (e.g., known drug or alcohol abuse or mental illness) that the investigator considered would have prevented the patient from complying with and completing the study protocol.
* Presence of any blood disorders that may interfere with HbA1c measurements (e.g., hemolytic anemia, sickle cell disease).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
blood sugar changes | 40 weeks
  Effects of Tirzepatide and Insulin Glargine on blood sugar changes in Patients With Type 2 Diabetes Mellitus
blood lipid changes | 40 weeks
  Effects of Tirzepatide and Insulin Glargine on blood lipid changes in Patients With Type 2 Diabetes Mellitus
Brain function | 40 weeks
  Effects of Tirzepatide and Insulin Glargine on brain function through VBM and ASL-fMRI in Patients With Type 2 Diabetes Mellitus.

SECONDARY OUTCOMES:
Body composition analysis | 40 weeks
  Effects of Tirzepatide and Insulin Glargine on body composition in Patients With Type 2 Diabetes Mellitus. A body composition analysis will assess the fat and muscle makeup of your body.
Inflammation factors, including adiponectin,leptin,IL-1,IL-6,IL-18,TNF-α,ghrelin,asprosin. | 40 weeks
  Effects of Tirzepatide on inflammation factors in Patients With Type 2 Diabetes Mellitus,after being intervened for 40 weeks,changes of Inflammation factors were observed, including adiponectin,leptin,IL-1,IL-6,IL-18,TNF-α,ghrelin,asprosin.

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Ma, Doctor, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China